CLINICAL TRIAL: NCT04712487
Title: Frequency and Characteristics of Low-grade Infections of the Intervertebral Discs
Brief Title: Low-grade Infections of the Intervertebral Discs
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EK1078/2018
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Disc Degeneration
Keywords: low-grade infection; intervertebral disc; spine; cutibacterium acnes; culture; herpes simplex; modic changes; CRP; histopathology; microbiology; oswestry disability index; neck disability index
MeSH Terms: conditions — Intervertebral Disc Degeneration; Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Routine discectomy: Patients undergoing routine spine surgery due to degenerative disease of the spine
  Interventions: Diagnostic Test: Microbiological culture, viral PCR, histopathological analysis

INTERVENTIONS:
Diagnostic Test: Microbiological culture, viral PCR, histopathological analysis — Intervertebral disc tissue was sent to the laboratory for further analysis:
  Microbiological culture: Detection of bacterial growth Viral PCR: Detection of Herpes-Simplex-Type 1 virus, Herpes-Simplex-Type 2 virus, Cytomegalovirus Histopathological analysis: Inflammation signs of disc tissue

SUMMARY:
The purpose of this prospective, observational study was to evaluate frequency and characteristics of low-grade infections of the intervertebral discs in an unselected real-life patient population undergoing surgery for degenerative pathologies of the spine.

DETAILED DESCRIPTION:
Low-grade infection of the intervertebral discs, causing disc degeneration and consecutive pain and disability is reported in literature. Microorganisms are also held responsible for Modic Changes of the vertebral bodies.

Patients underwent surgery for degenerative pathology of the spine independent of this study. After being informed about this study, all patients giving written informed consent who met eligibility requirements were included. Treatment of the patients was independent of this study. Intraoperative removed disc tissue was examined using microbiological culture, viral polymerase chain reaction (PCR), and histopathological analysis.

Other used data were demographic data (Gender, age), Modic Changes on MRI, preoperative Oswestry Disability Index (ODI), preoperative Neck Disability Index (NDI), and preoperative C-reactive protein (CRP).

Frequency of positive microbiological culture findings, viral PCR, and inflammation signs in histopathological analysis was described, and statistical analysis was performed to identify if any of the above mentioned parameters influences the frequency of positive microbiological culture and Modic Changes significant.

ELIGIBILITY:
Inclusion Criteria:

* Spine surgery including discectomy due to degenerative diseases
* Availability of removed disc tissue for further analysis

Exclusion Criteria:

* Signs of spondylodiscitis (clinical signs, inflammation parameters, radiological)
* Suspected or known tumor disease
* Traumatic fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Bacterial growth | 1 week (Time from surgery until final result of microbiological culture was available)
  Number of intervertebral discs with at least one positive microbiological culture result

SECONDARY OUTCOMES:
HSV-1 | 1 week (Time from surgery until final result of PCR was available)
  Number of intervertebral discs with at least one positive result for Herpes-Simplex-Virus type 1
HSV-2 | 1 week (Time from surgery until final result of PCR was available)
  Number of intervertebral discs with at least one positive result for Herpes-Simplex-Virus type 2
CMV | 1 week (Time from surgery until final result of PCR was available)
  Number of intervertebral discs with at least one positive result for Cytomegalovirus
MC 1 | Measured on preoperative MRI (maximum 3 months old)
  Positive Modic Change type 1 in the operated segment
MC 2 | Measured on preoperative MRI (maximum 3 months old)
  Positive Modic Change type 2 in the operated segment
MC 3 | Measured on preoperative MRI (maximum 3 months old)
  Positive Modic Change type 2 in the operated segment
ODI | Measured preoperative at hospital admission, i.e. 1-3 days before operation
  Oswestry Disability Index, measured only in case of lumbar spine surgery
NDI | Measured preoperative at hospital admission, i.e. 1-3 days before operation
  Neck Disability Index, measured only in case of cervical spine surgery
CRP | Measured preoperative at hospital admission, i.e. 1-3 days before operation
  C-reactive protein in mg/dl, measured as blood sample
Pathology | 1 week (Time from surgery until final result of histopathological analyzsis was available)
  Positive inflammation signs in histopathological analysis. Analyzed for each collected intervertebral disc

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Senker, MD, Principal Investigator — Kepler University Hospital
Locations (1):
- Department of Neurosurgery, Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iyer S, Louie PK, Nolte MT, Phillips FM. The Relationship Between Low-Grade Infection and Degenerative Disk Disease: A Review of Basic Science and Clinical Data. J Am Acad Orthop Surg. 2019 Jul 15;27(14):509-518. doi: 10.5435/JAAOS-D-18-00257. PMID 30575599
- [Background] Stirling A, Worthington T, Rafiq M, Lambert PA, Elliott TS. Association between sciatica and Propionibacterium acnes. Lancet. 2001 Jun 23;357(9273):2024-5. doi: 10.1016/S0140-6736(00)05109-6. No abstract available. PMID 11438138
- [Derived] Senker W, Aspalter S, Radl C, Pichler J, Doppler S, Weis S, Webersinke C, Wagner H, Hermann P, Aichholzer M, Aufschnaiter-Hiessbock K, Thomae W, Stroh N, Hauser T, Gruber A. Frequency and characteristics of bacterial and viral low-grade infections of the intervertebral discs: a prospective, observational study. J Orthop Traumatol. 2022 Mar 18;23(1):15. doi: 10.1186/s10195-022-00633-y. PMID 35303173